CLINICAL TRIAL: NCT05497622
Title: Quantitative Ultrasound Biomarkers to Assess Upper Trapezius Muscles in Patients With Chronic Neck Pain Before and After Osteopathic Manipulative Treatment
Brief Title: Quantitative Ultrasound Biomarkers to Assess Upper Trapezius Muscles in Patients With Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rocky Vista University, LLC (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #2022--095
Record Dates: First submitted 2022-08-01; First posted 2022-08-11 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Two groups will be used in the study to evaluate Quantitative Ultrasound Imaging (QUI) biomarkers and TART assessments.
  1. Healthy participants. Non-invasive quantitative ultrasound (B-mode image, ultrasound elastography), EMG, and osteopathic assessment (TART assessments) will be performed on the upper trapezius muscle in healthy controls one time at the time of the enrollment.
  2. Patients with chromic neck pain. Non-invasive quantitative ultrasound (B-mode ultrasound, ultrasound elastography), EMG, osteopathic assessment, and osteopathic manipulative treatment (OMT) of the upper trapezius muscle will be performed on participants with chronic neck pain 3 times. All ultrasound, EMG biomarkers and TART assessments will be collected before and after OMT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy participants (Experimental): Non-invasive quantitative ultrasound (B-mode image, ultrasound elastography), EMG, and osteopathic assessment (TART assessments) will be performed on the upper trapezius muscle in healthy participants one time at the time of the enrollment.
  Interventions: Diagnostic Test: Quantitative Ultrasound; Diagnostic Test: Osteopathic TART Assessment
- Patients with chronic neck pain (Experimental): Non-invasive quantitative ultrasound (B-mode ultrasound, ultrasound elastography), EMG, osteopathic assessment, and osteopathic manipulative treatment (OMT) of the upper trapezius muscle will be performed on participants with chronic neck pain 3 times. All ultrasound, EMG biomarkers and TART assessments will be collected before and after OMT.
  Interventions: Diagnostic Test: Quantitative Ultrasound; Diagnostic Test: Osteopathic TART Assessment; Procedure: Osteopathic Manipulation Treatment

INTERVENTIONS:
Diagnostic Test: Quantitative Ultrasound — Ultrasound assessment of Trapezius muscle
  Other Names: QUI
Diagnostic Test: Osteopathic TART Assessment — Evaluation of the 4 diagnostic criteria:
  1. Tissue Texture abnormality
  2. Asymmetry
  3. Restriction of Motion
  4. Tenderness
  Other Names: TART
Procedure: Osteopathic Manipulation Treatment — Use of manual techniques such as soft tissue stretching, resisted isometric stretches, fascial relaxation and counter strain.
  Other Names: OMT
  Arms: Patients with chronic neck pain

SUMMARY:
The goal of this study is to identify and develop multiparametric quantitative ultrasound imaging (QUI) biomarkers for assessing upper trapezius muscle with and without chronic neck pain and their response to treatment. This goal will be achieved by testing the underlying hypothesis that abnormal muscle tissue can be identified based on its physio-mechanical properties, and that changes in these properties can be used to guide and monitor treatment progress. Preliminary results have shown that biomarkers including muscle B-mode ultrasound echo-intensity, shear wave velocity, and longitudinal strain ratios associated with muscle tissue structure, mechanics, and function significantly differ between muscles in low back pain and neuromuscular disorders and normal muscles. This study will determine which biomarkers are best suited to differentiate abnormal muscle in chronic neck pain from healthy muscles and develop a quantitative objective program for chronic neck pain management.

DETAILED DESCRIPTION:
The main objective will be achieved through two aims:

Aim 1: Identify and develop quantitative biomarkers to distinguish structure, mechanics, function, and blood flow in abnormal muscles associated with chronic neck pain from normal muscles, correlated with clinical osteopathic assessments.

To determine the diagnostic performances of echo-intensity as a muscle structural biomarker, shear wave velocity and longitudinal strain ratio as muscle mechanics/function biomarkers, and color Doppler microvascular index as a muscle blood flow biomarker will be evaluated. These assessments will be evaluated in healthy subjects to test these quantitative biomarkers on upper trapezius muscle in the neck region to establish normal control values. To determine the clinical utility of these novel biomarkers, subjects with chronic neck pain will receive clinical osteopathic assessments over the neck region using conventional osteopathic examination with qualitative disease scoring by clinicians and subjective pain scales by subjects. The above quantitative biomarkers and qualitative osteopathic assessments of corresponding tissues with and without chronic neck pain will be analyzed using advanced ultrasound processing methods and statistical analyses.

Aim 2: Evaluate the abilities of quantitative biomarkers developed in Aim 1 to assess the responses of muscle tissue structure, mechanics, function, and blood flow to osteopathic manipulative treatment (OMT) for chronic neck pain.

To determine the prognostic performance of the QUI biomarkers developed in Aim 1 in predicting clinical response to OMT treatment, it will demonstrate that abnormal muscle tissue physio-mechanical properties to be directly linked to the pain of the patients. This trial will determine if improvement in abnormal biomarker values leads to improvement in subject's pain and osteopathic assessments. Subjects with chronic neck pain will be examined at intervals with biomarker measurements and osteopathic assessments. Image processing and statistical analysis will be used to determine the performance of the biomarkers in predicting response to treatment. the approach used in this study is supported by preliminary studies, which show how ultrasound biomarkers change following OMT, returning toward more normal muscle tissue mechanics.

This clinical trial will validate at least one clinically useful prognostic biomarker for chronic neck pain management, lay the foundation for further clinical research and treatment based on quantitative, reproducible, well-established methods, and lead to a large grant application.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the healthy participants include:

* Age 18 years and older;
* Healthy. No history of musculoskeletal conditions, such as severe pain, trauma, joint or spine surgery;
* Able to sign written informed consent,
* Tolerant to the osteopathic exam, and ultrasound.

Inclusion criteria for patients with chronic neck pain include:

* Age 18 years and older
* Having chronic neck pain persisting longer than 12 weeks, meeting TART criteria, diagnosed by an osteopathic physician;
* Able to sign written informed consent;
* Tolerant to the osteopathic exam, ultrasound, and OMT.

Exclusion Criteria:

Exclusion criteria for the healthy participants include:

* Under 18 years of age;
* Having a medical history of musculoskeletal conditions, joint and/or spine surgery, trauma;
* Employee of the study investigators;
* Being unable to competently consent or assent to participation (e.g., mentally disabled, demented, delusional, or a prisoner);
* Not tolerant to the osteopathic exam, ultrasound.

Exclusion criteria for patients with chronic neck pain include:

* Age < 18 years,
* Unable or unqualified to sign an informed consent,
* Unstable and/or late stage diseases,
* Not tolerant to the osteopathic exam, ultrasound, OMT.

There is no specific racial/ethnic background limitation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound diagnostic performance evaluation | Baseline, pre-intervention
  Evaluation for healthy participants and for patients with chronic neck pain. Changes in muscle B-mode ultrasound echo-intensity (arbitrary units), shear wave velocity (m/s), and longitudinal strain ratios (arbitrary units) will be recorded.
  Measured using ultrasound.
Ultrasound diagnostic performance evaluation | Immediately after the intervention
  Evaluation for patients with chronic neck pain. Changes in muscle B-mode ultrasound echo-intensity (arbitrary units), shear wave velocity (m/s), and longitudinal strain ratios (arbitrary units) will be recorded.
  Measured using ultrasound.

SECONDARY OUTCOMES:
Ultrasound echo-intensity | Baseline, pre-intervention
  Evaluation for healthy participants and for patients with chronic neck pain. Changes in muscle B-mode ultrasound echo-intensity (arbitrary units) will be recorded.
  Measured using ultrasound.
Ultrasound echo-intensity | Immediately after the intervention
  Evaluation for patients with chronic neck pain. Changes in muscle B-mode ultrasound echo-intensity (arbitrary units) will be recorded.
  Measured using ultrasound.
Ultrasound echo-intensity | Follow- up. Up to 18 weeks after procedure.
  Evaluation for patients with chronic neck pain. Changes in muscle B-mode ultrasound echo-intensity (arbitrary units) will be recorded.
  Measured using ultrasound.
Ultrasound shear wave velocity | Baseline, pre-intervention
  Evaluation for healthy participants and for patients with chronic neck pain. Changes in shear wave velocity (m/s), will be recorded. Measured using ultrasound.
Ultrasound shear wave velocity | Immediately after the intervention
  Evaluation for patients with chronic neck pain. Changes in shear wave velocity (m/s), will be recorded. Measured using ultrasound.
Ultrasound shear wave velocity | Follow- up. Up to 18 weeks after procedure.
  Evaluation for patients with chronic neck pain. Changes in shear wave velocity (m/s), will be recorded. Measured using ultrasound.
Ultrasound longitudinal strain ratios | Baseline, pre-intervention
  Evaluation for healthy participants and for patients with chronic neck pain. Changes in longitudinal strain ratios (arbitrary units) will be recorded. Measured using ultrasound.
Ultrasound longitudinal strain ratios | Immediately after the intervention
  Evaluation for patients with chronic neck pain. Changes in longitudinal strain ratios (arbitrary units) will be recorded. Measured using ultrasound.
Ultrasound longitudinal strain ratios | Follow- up. Up to 18 weeks after procedure.
  Evaluation for patients with chronic neck pain. Changes in longitudinal strain ratios (arbitrary units) will be recorded. Measured using ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Gao, MD, Principal Investigator — Rocky Vista University
Locations (1):
- Ultrasound Research Laboratory, Ivins, Utah, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be available with reasonable request to principal investigator.